CLINICAL TRIAL: NCT02309892
Title: A Phase I, Open Label, Dose Escalation Study of Immunoconjugate L-DOS47 in Combination With Pemetrexed/Carboplatin in Patients With Stage IV (TNM M1a and M1b) Recurrent or Metastatic NSCL Lung Cancer
Brief Title: A Dose Escalation Study of L-DOS47 in Recurrent or Metastatic Non-Squamous NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrolment - standard of care evolved over the duration of the study such that treatment regimen employed in the study was no longer current standard of care for first line resulting in recruitment challenges.
Sponsor: Helix BioPharma Corporation (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LDOS001
Record Dates: First submitted 2013-04-09; First posted 2014-12-05 (Estimated); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Neoplasms; Immunoconjugate; Tumor microenvironment alkalinization
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, dose escalation where patients are recruited into cohorts of escalating doses of L-DOS47 (0.59 up to 12.0 µg/kg) in combination with pemetrexed and carboplatin.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed and Carboplatin plus L-DOS47 (Experimental): Patients will be recruited into cohorts of L-DOS47 escalating doses, with a minimum of 3 and a maximum of 6 patients per cohort for the first and last two dosing cohorts, and a minimum of 1 and a maximum of 2 patients for the middle three dosing cohorts. The starting dose of L-DOS47 will be 0.59 µg/kg; further planned dose levels to be assessed are 0.78, 1.5, 3.0, 6.0, 9.0 and 12.0 µg/kg. The standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], respectively, to be administered in combination with L-DOS47, will remain constant across cohorts.
  Interventions: Drug: L-DOS47

INTERVENTIONS:
Drug: L-DOS47 — A treatment cycle will be 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle.

SUMMARY:
The primary purpose of this research study is to evaluate how safe, how well tolerated and how effective a range of doses of L-DOS47 in combination with standard doublet therapy of pemetrexed/carboplatin in patients with Stage IV (TNM M1a and M1b) recurrent or metastatic non-squamous Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
It is planned that patients will receive 4 cycles of combination treatment with L-DOS47 + pemetrexed/carboplatin. Patients who have not progressed following the 4 cycles of combination treatment and who have not experienced unacceptable toxicity will have the opportunity to continue to receive L-DOS47 treatment for as long as there is clinical benefit and it is well-tolerated, in the opinion of the Investigator, until disease progression. Patients who are unable to complete 4 cycles of L-DOS47 + pemetrexed/carboplatin combination treatment due to pemetrexed/carboplatin toxicity will have the opportunity to continue receiving L-DOS47 treatment following discontinuation of pemetrexed/carboplatin, for as long as there is clinical benefit and it is well-tolerated, in the opinion of the Investigator, until disease progression.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female patient ≥ 18 years of age
2. Histologically or cytologically confirmed non-squamous NSCLC
3. EGFR-mutation positive patients must have progressed on or had intolerance to an EGFR small molecule tyrosine kinase inhibitor
4. Patients whose tumors harbor an anaplastic lymphoma kinase (ALK) translocation must have progressed on or had intolerance to an ALK inhibitor;
5. No prior adjuvant chemotherapy within 1 year of the first treatment day if there is recurrent disease
6. At least 1 site of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and minimum life expectancy of ≥ 3 months
8. Adequate bone marrow, renal and liver function

Main Exclusion Criteria:

1. Histologic evidence of predominantly squamous cell NSCLC
2. Brain metastasis and/or leptomeningeal disease (known or suspected)
3. Peripheral neuropathy > CTCAE grade 1
4. Possibility of a curative local treatment (surgery and/or radiotherapy)
5. Previous chemotherapy except adjuvant treatment with progression of disease documented ≥ 12 months after end of adjuvant treatment
6. Having received treatment in another clinical study within the 30 days prior to commencing study treatment or having side effects of a prior study drug that are not recovered to grade ≤ 1 or baseline, except for alopecia
7. Concurrent chronic systemic immunotherapy, chemotherapy or hormone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Helix BioPharma corporate website — http://www.helixbiopharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were enrolled at three study sites in the United States from April 2014 to August 2019.
Pre-assignment Details: A total of 14 study subjects diagnosed with metastatic or recurrent non-small cell lung cancer (NSCLC) were enrolled to receive planned escalating doses of L-DOS47 (0.59 - 12.0 ug/kg) in combination with standard doses of carboplatin and pemetrexed.
Groups:
- L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 0.59 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 0.78 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 1.5 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 3.0 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 6.0 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 9.0 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 12.0 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
Period: Overall Study
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
Started | 3 | 6 | 1 | 1 | 1 | 2 | 0
Completed | 1 | 5 | 0 | 1 | 0 | 1 | 0
Not Completed | 2 | 1 | 1 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were no patients enrolled in cohort 7 (L-DOS47 12.0 ug/kg), as the study was concluded due to slow recruitment.
Groups:
- L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 0.78 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
- Total: Total of all reporting groups
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin | Total
Number analyzed (Participants) | 3 | 6 | 1 | 1 | 1 | 2 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 1 | 1 | 0 | 1 | 0 | 7
  >=65 years | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (3.00) | 62.8 (5.27) | 48 (0) | 56 (0) | 67 (0) | 65.5 (10.61) |  | 63.5 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 0 | 0 | 1 |  | 7
  Male | 2 | 2 | 0 | 1 | 1 | 1 |  | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 0 |  | 2
  White | 3 | 4 | 0 | 1 | 1 | 2 |  | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG performance status describes how daily living activities of the patient are affected by disease. ECOG of 0 means the patient is fully active without restriction. ECOG of 1 means the patient is restricted in physically strenuous activity but is able to carry out light work. The investigator assigned the ECOG score at baseline (i.e., before the patient started study treatment).
  Participants
    ECOG=0 | 1 | 3 | 0 | 0 | 0 | 0 |  | 4
    ECOG=1 | 2 | 3 | 1 | 1 | 1 | 2 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events as a Measure Safety and Tolerability of L-DOS47 in Combination Treatment With Pemetrexed/Carboplatin
Description: Beginning with the start of study treatment at Cycle 1 Day 1 up to the last study visit: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose which results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or, is a congenital anomaly/birth defect. Beginning with the AE reporting period at the start of study treatment at Cycle 1 Day 1 up to the last study visit;
Time Frame: Up to 12 weeks
Population: Any subject who has received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
Number analyzed (Participants) | 3 | 6 | 1 | 1 | 1 | 2 | 0
Participants
  Treatment emergent AEs | 3 | 6 | 1 | 1 | 1 | 2 |
  Treatment emergent AEs related to L-DOS47 | 2 | 5 | 0 | 0 | 0 | 0 |
  Treatment emergent SAEs | 0 | 3 | 0 | 1 | 1 | 1 |
  Treatment emergent SAEs related to L-DOS47 | 0 | 0 | 0 | 0 | 0 | 0 |

2. Primary Outcome: Number of Participants With Dose Limited Toxicities (DLTs) Related to L-DOS47 in Combination Treatment With Pemetrexed/Carboplatin.
Description: A DLT was defined as the occurrence of any of the following events (according to NCI CTCAE version 4.0) that are considered to be (possibly/probably/definitely) related to L-DOS47 and occurring within 21 days after commencing study treatment:
  * Haematological adverse events ≥ grade 4
  * Non-haematological adverse events ≥ grade 3
  * One instance each of any two unique grade 2 adverse events
Time Frame: Up to 21 days
Population: Any subject who has received all scheduled doses of L-DOS47 in Cycle 1; a DLT is assumed to have occurred if a patient does not receive all scheduled doses of L-DOS47 due to toxicity
Measure: Count of Participants; unit: Participants
Groups:
- L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin; L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin; L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin; L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin: Subjects were to receive a weekly dose 0.59 µg/kg of L-DOS47 by IV infusion in combination with standard of care doses of pemetrexed [500 mg/m2] and carboplatin [AUC6], where a treatment cycle was 21 days, with patients receiving L-DOS47 on cycle Days 1, 8, and 15 and pemetrexed/carboplatin on Day 1 of each treatment cycle for a total of four treatment cycles. Subjects had the option to continue on weekly doses of L-DOS47 for long as there was clinical benefit and well-tolerated.
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
Number analyzed (Participants) | 3 | 6 | 1 | 1 | 1 | 2 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 |

3. Primary Outcome: Maximum Tolerated Dose of L-DOS47 in Combination With Pemetrexed/Carboplatin
Description: Defined as the highest dose level at which ≤ 1 of 6 patients experiences a dose limiting toxicity (DLT) as assessed during the first treatment cycle. If no DLT are reported, it is assumed that the maximum tolerated dose of L-DOS47 in combination with pemetrexed/carboplatin was not reached.
Time Frame: 21 days
Population: Any subject who experienced a dose-limiting toxicity (DLT); a DLT is also assumed to have occurred if a patient does not receive all scheduled doses of L-DOS47 due to toxicity
Measure: Count of Participants; unit: Participants
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
Number analyzed (Participants) | 3 | 6 | 1 | 1 | 1 | 2 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 |

4. Secondary Outcome: Objective Response Rate of Patients Receiving the Combination Treatment According to RECIST 1.1
Description: Objective tumor response will be assessed according to RECIST version 1.1 in patients who have completed at least 2 cycles of study treatment and who have at least 1 post-treatment disease assessment; where complete response (CR) is the disappearance of all target lesions and partial response (PR) is at least a 30% reduction in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 12 weeks
Population: Efficacy-evaluable population includes those patients who have completed at least two cycles of study treatment and had at least one post-baseline tumor assessment. For patients with fewer than two cycles of study treatment, there had to be clear evidence of clinical progression. For patients to be evaluable for stable disease, the duration of stable disease must be at least 42 days from the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
Number analyzed (Participants) | 1 | 6 | 1 | 1 | 1 | 2 | 0
Participants
  Partial response | 1 | 3 | 0 | 1 | 0 | 0 |
  Stable disease | 0 | 1 | 1 | 0 | 0 | 2 |
  Progressive disease | 0 | 2 | 0 | 0 | 1 | 0 |

5. Secondary Outcome: Percentage of Patients Receiving a Sustained Clinical Benefit
Description: Defined as the percentage of patients who have achieved complete response, partial response, or stable disease following combination treatment with L-DOS47 + pemetrexed/carboplatin; where complete response (CR) is the disappearance of all target lesions, partial response (PR) is at least a 30% reduction in the sum of diameters of target lesions, taking as reference the baseline sum diameters, and stable disease (SD) is where neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD, at least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study).
Time Frame: Up to 12 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
Number analyzed (Participants) | 1 | 6 | 1 | 1 | 1 | 2 | 0
Participants | 1 | 4 | 1 | 1 | 0 | 2 |

ADVERSE EVENTS:
Time Frame: Adverse event (AE) reporting period commenced after initial dosing of pemetrexed premedication through 30-day post-last dose of study drug, up to 15 weeks, or longer for those patients who continue on additional treatment cycles. If an AE occurred before first dose of study drug, it would be considered a non-treatment emergent AE. All AEs were followed until resolution/stabilization while patient remained on-study.
Description: Once a patient was removed from study, events thought to be related to the study drug were followed until resolution/stabilization, unless, in the opinion of the investigator, event is unlikely to resolve due to the patient's underlying disease, or until the patient starts a new treatment regiment or is lost to follow-up.
Arm/Group | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/6 | 0/1 | 1/1 | 1/1 | 1/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 0/1 | 1/1 | 1/1 | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 1/1 | 1/1 | 1/1 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin (N=3) | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin (N=6) | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin (N=1) | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=1) | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=1) | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=2) | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=0)
nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-DOS47 0.59 ug/kg in Combination With Pemetrexed and Carboplatin (N=3) | L-DOS47 0.78 ug/kg in Combination With Pemetrexed and Carboplatin (N=6) | L-DOS47 1.5 ug/kg in Combination With Pemetrexed and Carboplatin (N=1) | L-DOS47 3.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=1) | L-DOS47 6.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=1) | L-DOS47 9.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=2) | L-DOS47 12.0 ug/kg in Combination With Pemetrexed and Carboplatin (N=0)
nausea (Gastrointestinal disorders) | 0 | 5 | 1 | 1 | 1 | 1 | 0
constipation (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
diarrhea (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
gastroesophageal reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
fatigue (General disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
oedema peripheral (General disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0
chest pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
pyrexia (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
weight fluctuation (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0
neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0
alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
hyperdrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
rash generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
neutrophil count decreased (Investigations) | 2 | 1 | 1 | 1 | 0 | 0 | 0
white blood cell count decreased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 0
platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0
alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
bone swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
neuropathy peripheral (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | NA
viral upper respiratory infection (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
defect conduction intraventricular (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Patient enrolment was halted at cohort 6 (9.0 ug/kg) due to slow recruitment and therefore, the seventh and highest dosing cohort (12 ug/kg) could not be completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02309892/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02309892/SAP_001.pdf